CLINICAL TRIAL: NCT04422912
Title: A Phase 1/2, Open-label, Safety and Dosing Study of Autologous CART Cells (Desmoglein 3 Chimeric Autoantibody Receptor T Cells [DSG3-CAART] or CD19-specific Chimeric Antigen Receptor T Cells [CABA-201]) in Subjects With Active, Pemphigus Vulgaris
Brief Title: A Phase 1/2, Open-label, Safety and Dosing Study of Autologous CART Cells (Desmoglein 3 Chimeric Autoantibody Receptor T Cells [DSG3-CAART] or CD19-specific Chimeric Antigen Receptor T Cells [CABA-201]) in Subjects With Active, Pemphigus Vulgaris (RESET-PV)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cabaletta Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAB-101
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pemphigus Vulgaris
Keywords: Pemphigus; Pemphigus Vulgaris; CAAR-T Therapy; CAR-T Therapy; Desmoglein 3; Cell Therapy; Autoimmune Disease; Autoimmunity; Skin Diseases, Vesiculobullous; Immunotherapy, Adoptive; Immune System Diseases; CABA-201; Anti-CD19 CAR-T therapy; Resecabtagene Autoleucel; Rese-cel
MeSH Terms: conditions — Pemphigus; Autoimmune Diseases; Skin Diseases, Vesiculobullous; Immune System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DSG3-CAART (Experimental): Single or multiple intravenous infusion(s) of DSG3-CAART at varying dose levels.
  This study is now closed to enrollment.
  Interventions: Biological: DSG3-CAART
- CABA-201 (Experimental): Infusion of CABA-201 with or without cyclophosphamide and fludarabine preconditioning, or with or without cyclophosphamide preconditioning.
  This sub-study is open to enrollment.
  Interventions: Biological: CABA-201

INTERVENTIONS:
Biological: DSG3-CAART — Intravenous infusions of DSG3-CAART alone at different doses and different fractionations, with or without intravenous immunoglobulin, cyclophosphamide, and/or fludarabine.
  Arms: DSG3-CAART
Biological: CABA-201 — Single intravenous infusion of CABA-201 at escalating doses, with or without preconditioning.
  Arms: CABA-201

SUMMARY:
A phase 1/2, open-label, safety and dosing study of autologous CART cells (desmoglein 3 chimeric autoantibody receptor T cells [DSG3-CAART] or CD19-specific Chimeric Antigen Receptor T cells [CABA-201]) in subjects with active, pemphigus vulgaris

DETAILED DESCRIPTION:
Pemphigus vulgaris (PV) is a B-cell mediated autoimmune disorder in which painful blisters are formed on the skin or mucosal membrane, including the mouth, nose, throat, eyelids, anus, and genitals.

This phase 1/2 study is being conducted in two parts. The first part is the main study conducted to find the maximum tolerated dose and optimal fractionated infusion schedule of an investigational cell therapy, DSG3-CAART, that can be given to patients with mucosal PV who are inadequately managed by standard therapies. This study is closed to enrollment.

The second part is a sub-study is being conducted to investigate if CABA-201, also called resecabtagene autoleucel, or "rese-cel", can be safely administered while achieving clinical responses without the need for preconditioning in mucosal-dominant PV (mPV) and mucocutaneous PV (mcPV) patients. This sub-study is open to enrollment.

DSG3-CAART or CABA-201 may potentially lead to complete and durable remission of disease.

ELIGIBILITY:
Inclusion Criteria for DSG3-CAART: Closed to enrollment

* Confirmed diagnosis of mPV by prior or screening biopsy and prior positive anti- DSG3 antibody ELISA
* mPV inadequately managed by at least one standard immunosuppressive therapies
* Active mPV at screening
* Anti-DSG3 antibody ELISA positive at screening

Inclusion Criteria for CABA-201 sub-study: Open to enrollment

* Age ≥18
* Confirmed diagnosis of PV by prior or screening biopsy and prior positive DSG3 ELISA, IIF, and/or DIF
* PV inadequately managed by at least one standard immunosuppressive therapy
* Active PV at screening
* DSG3 ELISA positive at screening

Exclusion Criteria:

* Active cutaneous lesions associated with PV that indicates mucocutaneous rather than mucosal-dominant disease
* Rituximab in last 12 months unless PV symptoms have recently worsened or anti-DSG3 antibody titers have recently increased
* Prednisone > 0.25mg/kg/day
* Other autoimmune disorder requiring immunosuppressive therapies
* Investigational treatment in last 3 months

Exclusion Criteria for CABA-201 sub-study

* Have paraneoplastic pemphigus or active malignancy (not including non-melanoma skin cancer) or malignancy diagnosed within the previous 5 years
* Have received rituximab or other anti-CD20 or anti-CD19 therapies in last 12 months unless anti-DSG3 antibody titers have recently increased or PV symptoms have recently worsened
* Prednisone > 0.25mg/kg/day
* Other autoimmune disorder requiring immunosuppressive therapies
* Treatment with any investigational agent within 4 weeks or 5 half-lives, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events, including Dose Limit Toxicity | 3 months
  Incidence of adverse events that are related to DSG3-CAART therapy
For CABA-201 Sub-study: To evaluate adverse events reported by subjects | Up to 28 days after CABA-201 infusion
  Incidence and severity of AEs

SECONDARY OUTCOMES:
Percent of CAAR-transduced cells | Baseline
  Percent of total cells for infusion that are CAAR-transduced cells by flow cytometry
Total DSG3-CAART positive cells | Baseline
  Total DSG3-CAART positive cells for each manufacturing run by flow cytometry
Cellular kinetics profile of DSG3-CAART | Up to 36 months
  Cellular kinetics profile of DSG3-CAART assessed by quantitative polymerase chain reaction
Change in DSG3 autoantibody titer | Up to 36 months
  Change in DSG3 autoantibody titer by ELISA compared to pre-infusion visit
Serologic remission | Up to 36 months
  Proportion of subjects achieving serologic remission, determined by negative DSG3 ELISA titer
Pemphigus Disease Area Index (PDAI) | Up to 36 months
  Change in PDAI compared to pre-infusion visit, scored on a 0-250 scale where a greater number represents more disease activity
Clinical remission: complete remission off therapy and complete remission on minimal therapy | Up to 36 months
  Proportion of subjects achieving complete remission, determined by a PDAI activity score of 0 for at least 2 months, either off therapy or on minimal therapy
Time to clinical remission and time to serologic remission | up to 36 months
  Time to clinical remission and time to serologic remission from the last infusion
Duration of clinical remission and duration of serologic remission | up to 36 months
  Duration of clinical remission and duration of serologic remission sustained after achieving the initial remission
For CABA-201 Sub-study: To evaluate adverse events reported by subjects | Up to 156 weeks after CABA-201 infusion
  Incidence and severity of AEs
For CABA-201 Sub-study: To characterize the pharmacodynamics (PD) | Up to 156 weeks
  Levels of B cells in the blood
For CABA-201 Sub-study: To characterize the pharmacokinetics (PK) | Up to 156 weeks
  Levels of CABA-201-positive T cells in the blood
For CABA-201 Sub-study: To evaluate autoantibody -related biomarkers | Up to 156 Weeks
  Levels of serum anti-DSG3 and anti-DSG1 antibodies
For CABA-201 Sub-study: To evaluate efficacy | Up to 156 Weeks
  Absolute and percent change in disease activity by Pemphigus Disease Area Index (PDAI)

CONTACTS AND LOCATIONS:
Overall Officials: Cabaletta Bio, Study Chair — Cabaletta Bio
Locations (13):
- United States (13):
  - Stanford University, Dept. of Dermatology, Redwood City, California
  - UC Davis, Dept. of Dermatology, Sacramento, California
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mount Sinai - Icahn School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of North Carolina, Department of Dermatology, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dept. of Dermatology, Dallas, Texas
  - MD Anderson Texas Medical Center, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No